CLINICAL TRIAL: NCT00482963
Title: A Pilot Study of the Pharmacokinetic Interactions Between the Hormonal Emergency Contraception, Plan B, and Efavirenz
Brief Title: A Study of the Drug Interactions Between a Hormonal Emergency Contraception and an HIV Medication
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Miriam Hospital (Other); University of Washington (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-1178
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections; Contraception; Pharmacokinetics
Keywords: HIV; Contraception; Antiretroviral agents; Pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — Levonorgestrel; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- levonorgestrel, efavirenz (Experimental): healthy HIV-negative women of reproductive age were given levonorgestrel, efavirenz
  Interventions: Drug: levonorgestrel, efavirenz

INTERVENTIONS:
Drug: levonorgestrel, efavirenz

SUMMARY:
The purpose of this study is to determine if blood levels of the hormonal emergency contraceptive agent, Plan B, are altered by concomitant use with the HIV medication, efavirenz.

DETAILED DESCRIPTION:
The use of hormonal contraceptive pills in women with HIV is complex due to potential interactions between these agents and HIV medications. HIV-infected women taking efavirenz have an even greater need for effective birth control as this medication may cause severe brain damage to a developing fetus. The use of an emergency contraceptive agent in cases of unprotected sex or condom failure can prevent pregnancy. This study seeks to establish that Plan B can be used effectively and safely in women taking efavirenz.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, HIV-1 seronegative women of child-bearing age.

Exclusion Criteria:

* Current use of hormonal contraception
* Pregnancy/Breast Feeding
* Post-menopausal status
* Obesity
* Hepatitis B or C
* Psychiatric illness
* Active Substance Abuse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The change in Plan B (levonorgestrel) Area under the Concentration Time Curve (AUC12) prior to and during steady state efavirenz | 12 hour pharmacokinetic study

SECONDARY OUTCOMES:
Pharmacokinetic parameters of levonorgestrel prior to and during steady state efavirenz | 12 hour pharmacokinetic study
Frequency of common levonorgestrel-associated adverse events prior to and during steady-state efavirenz | 3 weeks
Changes in liver function tests before and during efavirenz | 3 weeks
The efavirenz Area Under the Concentration Time Curve (AUC 24) in setting of levonorgestrel compared to historical controls | 12 hour pharmacokinetic study

CONTACTS AND LOCATIONS:
Overall Officials: Monica L Carten, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - The Miriam Hospital, Providence, Rhode Island